CLINICAL TRIAL: NCT06764901
Title: Scalable Technology for Online Prevention of Child Sexual Abuse (CSA) and CSA Materials - a Randomized Controlled Trial
Brief Title: Scalable Technology for Online Prevention of Child Sexual Abuse (CSA) and CSA Materials
Acronym: STOP-CSAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Universitat Internacional de Catalunya (Other); National Institute of Mental Health (NIMH) (NIH); University of Trás-os-Montes and Alto Douro (Other)
Responsible Party: Principal Investigator, Klaus Michael Beier, Prof. Dr. med. Dr. phil., Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8000186001; 101084719 (Other Grant/Funding Number: European Commission - Internal Security Fund (ISF-2021))
Record Dates: First submitted 2024-11-14; First posted 2025-01-09 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Sexual Behavior; Child Sexual Abuse Material (CSAM) Consumption; Behavioural Disorder; Behavior Problems; Online Behaviour
Keywords: Child Sexual Abuse Material (CSAM) consumption; CSAM; CSA; Pedophilia; Digital online intervention; CBT; Cognitive Behavioural Therapy; AI Assistant
MeSH Terms: conditions — Sexual Behavior; Mental Disorders; Pedophilia

STUDY DESIGN:
Intervention Model Description: * Randomized
  * Multi-centre
  * Open label
  * Parallel assignment
  * Superiority
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Waitlist (No Intervention): Control group: Waitlist.
- TCS Intervention (Experimental)
  Interventions: Behavioral: Online Therapy Chat Service (TCS)

INTERVENTIONS:
Behavioral: Online Therapy Chat Service (TCS) — Online Therapy Chat Service (TCS) based on CBT techniques from the Berlin Dissexuality Therapy (Beier, K. M. (2021). Pedophilia, hebephilia and sexual offending against children. The Berlin Dissexuality Therapy (BEDIT). Springer).
  Arms: TCS Intervention

SUMMARY:
1. Summary The STOP-CSAM Study is a two-armed randomized controlled trial of a non-pharmacological Therapy Chat Service for prevention of Child Sexual Abuse (CSA) and Child Sexual Abuse Materials (CSAM) in self-referred and self motivated patients with high frequent CSAM use and non-detected by the legal authorities.
2. Trial design This study is a prospective multicentred, stratified, parallel-group superiority study conducted in Germany, Czechia and Spain.
3. Background There has been a significant increase in child sexual abuse material (CSAM) on the internet in recent years. The use of CSAM is problematic especially because it creates a demand for and maintains contact child sexual abuse. Unfortunately, despite the significant increase in the number of CSAM users, limited resources are available for investigation and prosecution. Consequently, many users remain in the community, with neither intervention from the criminal justice system, nor the health system. The proposed study will examine whether a therapy chat service (TCS) intervention reduces the demand for, circulation and spread of CSAM in undetected offenders, as compared to a control group.
4. Methods The sample consists of individuals aged 18 years or older (expected N = 630), who have used CSAM in the prior two weeks and are seeking help voluntarily. Participants will be randomized to (1) a Therapy Chat Service (TCS) intervention or (2) a four-week waitlist (control group) followed by a TCS intervention. The TCS intervention group will receive four to six one-hour online therapy chat sessions over the period of four weeks, while the control group will remain on a waitlist for these four weeks before receiving the same TCS intervention. Assessments will be conducted at baseline (pre-intervention) and at 4-, 8-, 12- and 16-weeks post-intervention. The main objective of the study is to compare the effectiveness of TCS in the prevention of CSAM use within a sample of self-referred participants. The primary outcome is the significant decrease of CSAM consumption, which will be assessed by comparing self-reported severity and time spent using CSAM in the two weeks before the intervention and at four weeks following the intervention. Potential progress measures include time spent, severity and frequency of CSAM consumed. Psychological wellbeing and total sexual outlet will be also measured as secondary outcomes, other participant variables such as risk factors for CSAM consumption or sexual interests and therapeutic variables such as number of patient-therapist interactions, modules covered per session, common factors of psychotherapy, adverse effects of intervention and dropout rate will be also measured. Outcomes between groups will be compared following standard principles for RCTs.
5. Results The study will open for recruitment in October 2023, and data collection is expected to be completed by November 2024. The results for the primary outcomes are planned to be analysed by December 2024 and submitted for publication by the end of the project in March 2025.
6. Discussion The study will test whether the TCS intervention has a positive effect, not only in terms of reducing self-seeking potential sexual offenders' problematic sexual behaviours, but also on measures such as psychological wellbeing in CSAM users. Possible adverse effects of TCS intervention will also be assessed.

Recently, a similar trial called PRIOTAB-CBT, compared pre- and post-treatment outcome measures between a treatment group to a control group (Lätth et al., 2022). Results showed a significantly larger reduction in time spent using CSAM in the treatment group, in comparison to the control group. PRIOTAB-CBTh was a single-centre, single-blinded, psychological placebo-controlled RCT of an online cognitive behavioural psychotherapy. If the STOP-CSAM trial demonstrates that a TCS intervention reduces CSAM use, it could be an effective prevention strategy for sexual violence against children.

8. Funding European Commission - Internal Security Fund (ISF-2021).

ELIGIBILITY:
Inclusion Criteria:

* Adult participant (≥18 years);
* use of CSAM in the previous 2 weeks;
* English, German, Czech, Spanish or Portuguese speaker;
* voluntary participation and agreement with the terms of the study.

Exclusion Criteria:

* Having severe neuropsychiatric comorbidities (unstable psychotic disorder, organic brain damage, diminished intellectual capabilities, untreated drug or alcohol addiction);
* current inpatient psychiatric stays and/or any other current treatment for CSAM behaviour;
* CSA perpetration history (past or present);
* currently under a criminal investigation, proceeding, punishment or probation status for committing online or offline CSA or CSAM use

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
proportion of patients with a reduction in the severity or duration of CSAM use | At the end of waiting period and/or intervention, usually 4 to 6 weeks after onboarding and following up every two weeks up to 16 weeks after onboarding
  * Diminished severity or time spent in CSAM consumption:
    * Dichotomous outcome defined by a decrease of either a 50% or greater in time spent or of one level or greater of severity of the consumed materials, comparing week 1 and week 4.
    * Primary outcome assessment:
  * Severity (self-reported):
    o Adapted version of COPINE scale (Merdian et al., 2013):
  * Time (self-reported):
    * How much time did you spend in total using these materials during the last two weeks? (hh:mm)

SECONDARY OUTCOMES:
Frequency of CSAM consumption (self-reported) | every 2 weeks for 16 weeks after onboarding
  How often have you used these materials during the last two weeks?
  * Never
  * Once
  * Once/twice a week (2/4 times during last two weeks)
  * Several times a week (more than four times during last two weeks)
  * Every day
Increased mental wellbeing (composite) | comparing week 1 and week 4
  Dichotomous outcome defined by an increase of a 10% or greater in mental wellbeing
  o Mental wellbeing (self-reported):
  ● Measured with the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS; Tennant et al., 2007).
Total sexual outlet (self-reported) | every 2 weeks for 16 weeks after onboarding
  * How many orgasms did you achieve during the last week?
  * How many of these by masturbation?
  * How many of these by sexual interaction with other people?

CONTACTS AND LOCATIONS:
Locations (2):
- Charite - Universitätsmedizin Berlin, Berlin, Germany
- UIC, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes